CLINICAL TRIAL: NCT01096472
Title: Phase IIa, Two-center, Randomized, Double Blind Study With Parallel Groups to Evaluate the Anti-mycotic and Anti-inflammatory Efficacy of Topical Combinational Product LAS 41003 Versus Corresponding Mono-substances in Patients With Inflammatory Tinea Pedis
Brief Title: Efficacy and Safety of LAS41003 in the Treatment of Inflammatory Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 552 000-0919; 2009-016626-14 (EudraCT Number)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2010-11

CONDITIONS: Tinea Pedis
Keywords: Tinea pedis
MeSH Terms: conditions — Tinea Pedis | interventions — octenidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS41003 (Experimental): Once daily
  Interventions: Drug: LAS41003
- LAS189962 (Active Comparator): Once daily
  Interventions: Drug: LAS189962
- LAS189961 (Active Comparator): Once daily
  Interventions: Drug: LAS189961

INTERVENTIONS:
Drug: LAS41003 — Once daily
  Arms: LAS41003
Drug: LAS189961 — Once daily
  Arms: LAS189961
Drug: LAS189962 — Once daily
  Arms: LAS189962

SUMMARY:
The aim of this study is to determine the efficacy and safety of a topical application of the combinational cream LAS41003 compared to application of its mono-substances after once daily treatment in patients with inflammatory tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* presence of tinea pedis caused by dermatophytes on one or both feet, characterized by physician's global assessment score of 2 ("notable signs and symptoms exist") or 3 ("prominent signs and symptoms exist") at baseline;
* the physical examination must be without other disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the study;
* female volunteers of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 % per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices [IUDs], sexual abstinence or vasectomized partner;
* patients must be willing and able to comply with the requirements of the trial protocol;
* written informed consent obtained.

Exclusion Criteria:

* patients with hyperkeratotic chronic plantar tinea pedis (moccasin type);
* receiving systemic therapy with cytotoxic or immunosuppressive drugs either concurrently or within 12 weeks before the baseline visit;
* oral antifungal therapies within three months before study entry (8 months for oral terbinafine), systemic antibiotic or corticosteroid treatment, topical corticosteroids within 30 days before study entry;
* patients with diabetes;
* patients with compromised circulation;
* evidence of drug or alcohol abuse;
* pregnancy or nursing;
* symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before the treatment phase and during the study;
* participation in the treatment phase of another clinical study within the last four weeks prior to the first administration of investigational drug in this study;
* known allergic reactions to components of the study preparations, hypersensitivity against cetylstearyl alcohol;
* treatment with systemic or locally acting medications which might counter or influence the study aim within two weeks before the treatment phase of the study (e.g. glucocorticosteroids);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Clinical assessment scores and mycological status of fungi (KOH test and mycological culture) | 2 weeks

SECONDARY OUTCOMES:
Physicians assessment of signs and symptoms (erythema, scaling, vesicles, pustules, crusting, fissuring and maceration) | 2 weeks
  Percentage of locla skin reactions, AEs
Local skin reactions, AEs | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (2):
- Germany (2):
  - Investigational Site #2, Berlin
  - Investigational Site #1, Hamburg